CLINICAL TRIAL: NCT04482790
Title: Restoring Black Triangle With Bioclear Matrix and Injection Molding Technique Versus Celluloid Conventional Matrix Method: A Randomized Clinical Trial
Brief Title: Restoring Black Triangle With Bioclear Matrix Versus Celluloid Conventional Matrix Method
Acronym: RBBCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Omar Tawfik Hussien, Assistant lecturer in conservative department of faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-8-23
Record Dates: First submitted 2020-03-22; First posted 2020-07-23 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Gingival Black Triangle
Keywords: black triangle; bio-clear cervical matrix; dental esthetics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional celluloid matrix (Active Comparator): Conventional celluloid matrix technique in management of black triangle
  Interventions: Procedure: Conventional celluloid matrix technique in management of black triangle
- Bioclear cervical matrix (Experimental): Bioclear cervical matrix with injection molding technique in management of black triangle
  Interventions: Procedure: Bioclear cervical matrix with injection molding technique

INTERVENTIONS:
Procedure: Conventional celluloid matrix technique in management of black triangle — conventional restorative technique in management of black triangle
  Arms: Conventional celluloid matrix
Procedure: Bioclear cervical matrix with injection molding technique — New restorative technique in management of black triangle restorative papilla regeneration
  Arms: Bioclear cervical matrix

SUMMARY:
Assessment of bioclear matrix and injection molding technique against conventional celluloid matrix technique in management of black triangle.

DETAILED DESCRIPTION:
Patients with black triangle defect in anterior teeth (Cl I and Cl II according to Nordland and Tarnow classification) managed by Bioclear matrix with injection molding technique and conventional celluloid matrix technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the trial must comply with all of the following:

  * Cl I and cl II according to Nordland and Tarnow classification
  * Good oral hygiene
  * Good general health
  * Cooperative patient
  * Subjects who signed the informed consent
  * Patient compliance

Exclusion Criteria:

* Cl III according to Nordland and Tarnow classification
* Uncontrolled parafunction.
* Insufficient oral hygiene
* Periodontal and gingival diseases
* Pregnant and nursing
* Disabilities
* Systemic disease or severe medical complications
* Lack of compliance

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Esthetic evaluation | 12 months
  Scoring system according to World Dental Federation (FDI) criteria

SECONDARY OUTCOMES:
Marginal adaptation | 12 months
  Scoring system according to FDI criteria from one to five one represents very good clinically restoration & five represents poor clinically restoration

OTHER OUTCOMES:
Phonetics | 12 months
  Visual Analogue Scale (VAS) from zero to ten ,zero represents none & ten represent sever
Food impaction | 12 months
  Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Aya O Hussien, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Hussien AOT, Ibrahim SH, Essa MES, Hafez RM. Restoring black triangle with bioclear matrix versus conventional celluloid matrix method: a randomized clinical trial. BMC Oral Health. 2023 Jun 17;23(1):402. doi: 10.1186/s12903-023-03102-y. PMID 37330484